CLINICAL TRIAL: NCT01174641
Title: A Randomised Double-blind Test of TMS Intervention on Unilateral Neglect
Brief Title: Test of Trans-cranial Magnetic Stimulation (TMS) Intervention on Unilateral Neglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: The Stroke Association, United Kingdom (Other)
Responsible Party: Dr Brendan Laverty, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSA 2010/3
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Stroke
Keywords: unilateral neglect; TMS intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMS intervention (Experimental): Trans-cranial magnetic stimulation will be applied at a 1Hz rate for 20min over the ipsilesional posterior parietal cortex of patients showing left neglect after a right hemisphere stroke
  Interventions: Other: trans-cranial magnetic stimulation
- Placebo TMS (Placebo Comparator): 1 Hz trans-cranial magnetic stimulation will be applied over the vertex
  Interventions: Other: trans-cranial magnetic stimulation

INTERVENTIONS:
Other: trans-cranial magnetic stimulation — 1 Hz trans-cranial magnetic stimulation will be applied for 20min at 60% motor threshold over the vertex
  Arms: Placebo TMS
Other: trans-cranial magnetic stimulation — trans-cranial magnetic stimulation will be applied at 1Hz for 20 min over the ipsilesional posterior parietal cortex of stroke patients with unilateral neglect
  Arms: TMS intervention

SUMMARY:
Problems in attention can affect around 40% of stroke survivors and are associated with poor recovery of function. This project will provide the largest scale and most detailed examination to date of whether problems in attention after stroke can be remediated through direct brain stimulation. In Part 1 of the project the investigators will use two forms of direct brain stimulation (neural inhibition) to try and balance activity across the two sides of the brain following a stroke to one side. The investigators will assess whether each form of stimulation leads to an improvement in attentional functions, as well as to wider improvements in other cognitive abilities and to activities of everyday living. Performance will be tested immediately post remediation and on longer-term follow-up, and performance of the two intervention groups will be assessed against data the investigators have collected from a large-scale screen of cognitive impairments and recovery of function under standard treatment conditions. In Part 2 of the project the investigators will take the most promising intervention from Part 1 and the investigators will use magnetic resonance imaging (MRI) to determine the brain changes that are linked to the recovery of attentional functions. The investigators will test whether recovery is linked to a change in the balance of activation within the two hemispheres of the brain, and whether there are associated structural changes in cortical tissue and fibre tracts. The project will evaluate whether neural inhibition can improve attentional functions in particular, and cognitive abilities and everyday activities more generally, in stroke survivors. It will also provide novel information on how recovery of function comes about within the brain.

ELIGIBILITY:
Inclusion Criteria:

* presence of left unilateral neglect after right hemisphere stroke

Exclusion Criteria:

* presence of epilepsy/family history of epilepsy
* insufficient comprehension to follow instructions

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Standardised measure of visual neglect | 9 months
  A measure of unilateral neglect will be used

SECONDARY OUTCOMES:
measure of working memory | 9 months
  a standardised measure of working memory from the Birmingham University Cognitive Screen (www.bucs.bham.ac.uk)

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Humphreys, PhD, Principal Investigator — University of Birmingham
Locations (1):
- Queen Elizabeth Hospital, Birmingham, West Midlands, United Kingdom